CLINICAL TRIAL: NCT07178678
Title: A Phase II, Blinded, Randomized, Placebo-controlled Study to Evaluate the Safety and Efficacy of NeuroEPO in Subjects With Mild to Moderate Alzheimer's Disease Who Are Receiving Standard of Care Treatment
Brief Title: Evaluation of the Safety and Efficacy of NeuroEPO in Subjects With Mild to Moderate Alzheimer's Disease
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Center of Molecular Immunology, Cuba (Other)
Responsible Party: Principal Investigator, Andrew Kirk, Principal Investigator, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBIRD.NeuroEPO.20210803
Record Dates: First submitted 2024-11-25; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Mild Alzheimer's Disease; Moderate Alzheimer's Disease
Keywords: Alzheimer's Disease; NeuroEPO; EPO; ADAS-cog13

STUDY DESIGN:
Intervention Model Description: One group will receive NeuroEPO and one group will receive a placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NeuroEPO + standard of care (Experimental): NeuroEPO + standard of care for Alzheimer's Disease
  Interventions: Drug: NeuroEPO
- Placebo + standard of care (Placebo Comparator): Placebo + standard of care for Alzheimer's disease
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NeuroEPO — 0.5 mg of NeuroEPO will be administered intranasally three times a week for 52 weeks.
  Arms: NeuroEPO + standard of care
Drug: Placebo — 250 µL of placebo will be administered to intranasally to each nostril three times a week for 52 weeks.
  Arms: Placebo + standard of care

SUMMARY:
The goal of this clinical trial is to test if NeuroEPO improves or maintains cognition in adults with mild to moderate Alzheimer's Disease using a cannula attached to a syringe for delivery. It will also learn the safety of NeuroEPO. The main questions it aims to answer are:

Does NeuroEPO lower or maintain a person's cognition who has been diagnosed with Alzheimer's Disease? What medical problems do participants have when taking NeuroEPO?

Researchers will compare NeuroEPO to a placebo (a look-alike substance that contains no drug) to see if NeuroEPO works to treat Alzheimer's Disease.

Participants will:

Take NeuroEPO or a placebo three times a week for one year Visit the clinic to determine eligibility, for cognitive testing and blood tests at the start and end of the trial and at 1, 2, 6 and 12 months for check ups and blood collection

DETAILED DESCRIPTION:
The objective of the trial will be to assess the safety and efficacy of NeuroEPO plus standard of care treatment in participants with mild to moderate AD when delivered with a cannula attached to a syringe. A previous Phase II-III clinical trial in Cuba showed excellent safety and efficacy of NeuroEPO compared to no treatment in mild to moderate AD patients. In this clinical trial, NeuroEPO was administered intranasally with an insulin syringe. In the proposed phase II clinical trial, we will assess the safety and efficacy of 0.5 mg of NeuroEPO administered intranasally using a cannula attached to a syringe while the participant is in the Kaiteki position. Participants will be divided into two cohorts, involving 60 NeuroEPO-treated, and 30 placebo-treated participants for a total of 90 participants. NeuroEPO or the placebo will be administered three times a week for 52 weeks. An updated ADAScog test (ADAScog13) will be used as the primary outcome. The ADAScog13 test will be administered along with the other cognitive tests, Global Deterioration Scale (GDS), the Clinical Dementia Rating (CDR) the Mini Mental State Examination (MMSE), Alzheimer's Disease Co-operative Study Activities of Daily Living (ADCS-ADL), Neuropsychiatric Inventory Questionnaire (NPI-Q), Quality of Life in Alzheimer's Disease (QoL-AD) prior to starting treatment and one year after treatment. β-amyloid, phosphoTau, and ApoE biomarkers and the additional neuropsychological tests will be used as secondary outcomes. Labs, vitals and adverse events will be collected prior to the start of the trial, at 1, 3, 6, and 12 months to monitor for safety. Participants who consent to MRI and/or PET will be administered MRI and PET scans twice in the trial, once when the trial participant commences the trial and once when they conclude the trial. At 12 months final evaluations will be collected for cognitive tests and for those participants who consented to MRI and/or PET a second MRI and/or PET scan will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 50 years of age, to reflect the population that will be treated and to avoid younger populations who may be suffering dementia from a cause other than Alzheimer's Disease.
* Patients with Global Deterioration Scale (GDS) between 3 to 5 points (inclusive).
* Clinical Dementia Rating (CDR) - GS score 1-2 at screening.
* Patients with permeable airways.
* Patients (or caregiver, if the patient cannot) grant consent to participate in the study by signing the informed consent form.
* Patient with caregiver is physically and mentally willing to collaborate with the investigation.
* Mini-Mental State Examination (MMSE) score between 14 and 26 (inclusive) at screening

Exclusion Criteria:

* Evident mental disability or other limitation that prevents the patient or caregiver from administering the study evaluations.
* Patients with neurological symptoms or signs that suggest another cause of dementia.
* Skull trauma or recent intracranial surgery.
* Known clotting disorders.
* Use of anticoagulants, a medication to prevent harmful blood clots (warfarin, heparin or NOAC).
* Patients where coexistence of another disease or condition that may lead to significant disability (cancer, septic embolism, endocarditis, myeloproliferative disease, creatinine> 3 mg / dl (265µmol / L), hyperkalemia > 5.0 mmol / L, chronic/severe liver or kidney or heart disorders.
* Patients with a history of hypersensitivity to rhEPO.
* Patients with known allergy to any ingredients of the product.
* Patients who present nasal irritation (sneezing) or a runny nose before starting treatment.
* Patients who present asthma attack at the beginning of the treatment.
* Patients receiving treatment with AChE-I or Memantine who are not stable for 12-weeks prior to screening.
* Patients receiving treatment with psychoactive that can compromise the clinical trial results or neuropsychological tests.
* Patients with a history of alcoholism and/or drug dependence.
* Patients with chronic rhinosinusitis.
* Have a history of abnormal nasal or sinus symptoms.
* Have prior skull fracture or abnormality (nasal defect, deviated septum).
* Have recent nasal trauma (fracture in the last 2 months).
* Have any prior sinus or nose surgery (rhinoplasty).
* Have known bleeding problem (low platelets-thrombocytopenia), recurrent nose bleeds (>3 year).
* Have acute inflammation inside the nose.
* Congenital cranial facial disorders.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale - Cognitive (ADAS-cog13) | This test will be done prior to the start of treatment and at the end of treatment at 52 weeks
  The ADAS-cog13 is a brief battery of cognitive tests that assesses learning and memory, language production, language comprehension, constructional praxis, ideational praxis, and orientation. The ADAS-Cog is an in-person examiner-administered, structured scale that evaluates memory (word recall, word recognition), reasoning (following commands), language (naming, comprehension), orientation, ideational praxis (placing letter in envelope) and constructional praxis (copying geometric designs). Ratings of spoken language, language comprehension, word finding difficulty, and ability to remember test instructions are also obtained. The ADAS-cog13 scale is scored from 0-85, with higher scores indicating a worse outcome.

SECONDARY OUTCOMES:
Clinical Dementia Rating scale Sum of Boxes (CDR-SB) | This test will be done prior to the start of treatment and at the end of treatment at 52 weeks
  The CDR-SB describes five degrees of impairment in performance on each of six categories of cognitive functioning including memory, orientation, judgement, problem solving, community affairs, home and hobbies, and personal care. The CDR-SB scale is scored from 0-18, with higher scores indicating a worse outcome.
Mini-Mental State Exam (MMSE) | This test will be done prior to the start of treatment and at the end of treatment at 52 weeks
  The MMSE is a brief, frequently used screening instrument for AD drug studies. The MMSE scale evaluates orientation, memory, attention, concentration, naming, repetition, comprehension, ability to create a sentence, and to copy two overlapping pentagons. The MMSE scale is scored from 0-30, with lower scores indicating a worse outcome.
Neuropsychiatric inventory (NPI) | This test will be done prior to the start of treatment and at the end of treatment at 52 weeks
  The NPI is a well-validated, reliable, multi-item instrument to assess psychopathology in AD based on an interview with a caregiver or qualified study partner (defined in this study as having direct contact 10 hours/week). It evaluates both the frequency and severity of delusions, hallucinations, dysphoria, anxiety, agitation/aggression, euphoria, disinhibition irritability, lability, apathy, and aberrant motor behavior. The NPI scale is scored from 0-5, with lower scores indicating a worse outcome.
Alzheimer's Disease Cooperative Study - Activities of daily living (ADCS-ADL). | This test will be done prior to the start of treatment and at the end of treatment at 52 weeks
  Based on an interview with a caregiver or qualified partner, a participant is rated on his/her ability to carry out ten complex activities of daily living. The ADCS-ADL scale is scored from 0-78, with lower scores indicating a worse outcome.
Quality of Life in Alzheimer's disease (QoL-AD). | This test will be done prior to the start of treatment and at the end of treatment at 52 weeks
  The QoL-AD scale was developed by Logsdon et al. The QoL-AD is comprised of 13 items (physical health, energy, mood, living situation, memory, family, marriage, friends, self, ability to do chores, ability to do things for fun, money and life as a whole). Response options include 1 (poor), 2 (fair), 3 (good) and 4 (excellent), for a total score of 13-52, with higher scores indicating better QoL.
Blood analysis of phosphoTau (pTau) | This test will be done prior to the start of treatment and at the end of treatment at 52 weeks
  Measures biomarkers p-tau181 and p-tau217 in serum.
whole brain volume MRI (vMRI) | The scan will be done prior to the start of treatment and at the end of treatment at 52 weeks
  Alzheimer's disease (AD) is associated with excess whole brain volume loss, and progressive cognitive impairment. This is an optional scan.
Global Dementia Scale (GDS) | This test will be given prior to the start of treatment and at the end of treatment at 52 weeks.
  GDS is used as a screening tool that helps healthcare professionals assess the progression of a patient's dementia. The GDS is scored from 0-15, with higher scores indicating a worse outcome.
Blood analysis of Amyloid (Aβ1-42/Aβ1-40 ratio) | This test will be be done prior to treatment and at the end of treatment at 52 weeks.
  Serum detection of amyloid-beta

OTHER OUTCOMES:
Amyloid-PET (Vizamyl) | This test will be done prior to the start of treatment and at the end of treatment at 52 weeks
  Vizamyl conjugated to the isotope fluoride-18 (Vizamyl - F-18) (PET probe), is radioactive diagnostic agent indicated for Positron Emission Tomography (PET) imaging of the brain to estimate β-amyloid neuritic plaque density in adult patients with cognitive impairment who are being evaluated for Alzheimer's disease (AD). This is an optional scan.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: Undecided